CLINICAL TRIAL: NCT02619721
Title: Clinical Trial of Sacral Neuromodulation for Treatment of Refractory Overactive Bladder (OAB)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PINS-016
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-03

CONDITIONS: Refractory Overactive Bladder
Keywords: PINS SNS OAB
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Sacral Neuromodulation is on (Experimental): Sacral Neuromodulation is on as soon as implantation
  Interventions: Device: PINS SNS
- Sacral Neuromodulation is off (Placebo Comparator): Sacral Neuromodulation is off after implantation
  Interventions: Device: PINS SNS

INTERVENTIONS:
Device: PINS SNS

SUMMARY:
Evaluate the long-term clinical effectiveness and safety of the PINS Sacral Neuromodulation to patients with refractory Overactive Bladder.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 16 years OAB and/or OAB symptoms Refractory to standard medical therapy 100ml bladder capacity with normal upper urinary tract Good surgical candidate Able to complete study documentation and return for followup evaluation

Exclusion Criteria:

* Neurological conditions Stress urinary incontinence OAB symptoms caused by urinary tract infections

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-11 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Changes in voiding frequency from baseline to the voiding frequency evaluvation period 6 month | 6 month of stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China